CLINICAL TRIAL: NCT07328152
Title: CoMbination of Data From European Cohorts as Part of the European MORPHEUS Project [HORIZON-HLTH-2022-11-01] - "MC-MORPHEUS".
Acronym: MC-MORPHEUS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0090 - MC-MORPHEUS
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism; pulmonary embolism; Anticoagulant; deep vein thrombosis
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Combine clinical, biological and morphological data from 14 French and European cohorts into a single database.

DETAILED DESCRIPTION:
The MORPHEUS project is an international translational research programme selected and funded by the European call for proposals HORIZON-HLTH-2022-TOOL-11-01. This programme is coordinated by France (Brest University Hospital, INNOVTE, Inserm). This programme brings together all scientific disciplines and involves eight European countries: France, the Netherlands, Spain, Germany, Switzerland, Poland, Sweden and Denmark.

Based on quantitative and qualitative approaches, the MORPHEUS project will combine clinical, biological and morphological biomarkers (precision medicine: based on systematic literature reviews and cohort fusion) and socio-anthropological markers (personalised medicine: socio-anthropological interviews) in a risk prediction tool integrated into a shared medical decision-making process to aid therapeutic decision-making (duration and treatment modalities). The objective is to validate a time-dependent, multi-level tool integrated into a shared medical decision-making process to optimise long-term treatment of unprovoked venous thromboembolic disease (VTED) in a randomised stepped wedge cluster trial.

MC-MORPHEUS is a key phase of the MORPHEUS project aimed at identifying discriminatory biomarkers predictive of risk (thromboembolic recurrence, bleeding, mortality) that will form the basis of the MORPHEUS project's prediction tool.

The aim of the 'MC-MORPHEUS' project is therefore to combine, in a single database, clinical, biological and morphological data from European cohort databases of patients with VTE who have been monitored over several months and years. This combination of European cohort databases will increase the chances of identifying discriminating clinical, biological and morphological biomarkers for risk prediction. The identified and selected biomarkers will then be incorporated into the risk prediction tool, which will be validated in the ETHER cluster study of the MORPHEUS programme.

ELIGIBILITY:
Inclusion Criteria:

* Cohorts led by members of the European MORPHEUS project consortium European MORPHEUS project

Exclusion Criteria:

* Lack of consent in cohorts

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with MVTE who participated in one of the 14 French or European cohorts
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Consistency between merged data and initial data from each cohort | Processing of data from the fourth quarter of 2024 to the third quarter of 2025.
  The primary outcome is the consistency between the merged dataset and the original data from each cohort, assessed by comparing key variables across sources to ensure data integrity and accuracy. Consistency will be defined as the absence of significant discrepancies in predefined variables, such as demographic characteristics, baseline measures, and primary endpoints.

SECONDARY OUTCOMES:
Risk of thromboembolic recurrence | 20 YEARS
Risk of hemorrhagic complications | 20 YEARS
Risk of death | 20 YEARS

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement